CLINICAL TRIAL: NCT05609799
Title: The Distribution of Leucocyte Subsets in Healthy Danish Females of Reproductive Age
Brief Title: Distribution of Immune Cells Subsets in Healthy Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Caroline Nørgaard-Pedersen, dr.med., Aalborg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CNPOBC2020b
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2022-11

CONDITIONS: Healthy
Keywords: immune system
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: One group of healthy females. A blood sample is collected in the luteal phase; parts are saved for a biobank for future studies and parts are analyzed immediately for leucocyte subsets. This group will serve as a reference to other studies on (immunological) diseases in women of reproductive age.
Masking Description: No treatment intervention, only a blood sample is collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy females (Other): One blood sample is collected on healthy females in reproductive age. The sample will be analyzed for volumen of leucocyte subsets.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Quantifying the volume of leucocyte subsets: NK-cells, B-cells, and T-cell subsets, including Treg, Th1, Th2 and Th17 in EDTA

SUMMARY:
This study aims to evaluate the distribution of different lymphocyte subsets and other immune biomarkers in peripheral blood in healthy Danish females of reproductive age and to make a research biobank for future research. This data will serve as a reference to an ongoing study as well as future studies investigating the impact of the immune system on diseases affecting females in reproductive age.

DETAILED DESCRIPTION:
A blood sample will be collected from 37 healthy Danish females of reproductive age; part of material will be analysed immediately and part of it will be stored in a research biobank for future research. The samples are collected by clinicians at the Department of Gynaecology at Aalborg University Hospital (AaUH), and these samples are on the same day delivered to at the Department of Clinical Biochemistry (DCB) and Department of Clinical Immunology (DCI) at AaUH, that will perform the sample analyses. The DCI will store the biobank material.

The blood samples will be collected in EDTA-, citrate- and heparin-stabilised tubes. A white blood cell differential count, progesterone level measurement, and the leukocyte subset analysis will be performed by personnel at the DCB and DCI at AaUH.

Serum-progesterone level will be measured on the same day or the day before the blood samples for immunology testing and biobank is collected to ensure that the participant has ovulated and is in the luteal phase. Only blood samples with a serum progesterone level >20 nmol/l will be accepted for the study and included in the biobank. The result of the serum-progesterone measurement may come after the immunology analyses have started, but if the progesterone level is <20 nmol/l, further analyses will be cancelled, and the biobank material will be destroyed.

The white blood cell differential count (WBC) will be obtained from the Sysmex XN-1000 blood analyser. The analysis for NK-cells, B-cells, and T-cell subsets, including Treg, Th1, Th2 and Th17 in EDTA stabilised samples will be performed by the DCI on a flow cytometer using antibodies specific for surface markers that are exclusive for each leukocyte subset.

Blood for the research biobank comprises the remaining tubes. The serum and plasma in these three tubes will after immediate centrifugation be aliquoted and stored in tubes at -80 C in a locked freezer.

ELIGIBILITY:
Inclusion Criteria:

* - Healthy women of fertile age (18-41 years) with a regular menstrual cycle (22-35 days) who are in the luteal phase of their menstrual cycle at the time collecting the blood sample (day 20 to 28 of cycle and serum progesterone > 20 nmol/l at the day of blood sample). The group should consist of an approximately 1:1 ratio of women with ≥1 previous liveborn child and women with no previous pregnancy.

Exclusion Criteria:

* < 18 years old or >41 years old
* History of ≥1 known pregnancy loss including both spontaneous and missed abortions. An induced abortion is accepted if it was performed more than 2 years before study participation.
* Pregnancy within last 6 months
* Treatment with drugs acting on the immune system or hormonal contraceptive drugs either acting systemically or locally (intrauterine device releasing progesterone).
* Known disease with influence on the immune system and/or endocrine system
* Previously received a blood transfusion

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Volume of NK cells (CD56dim) | lutheal phase, day 20-28 in the menstrual cycle. The sample is collected at 9-10 AM and analysis is initiated within 60min.
  CD3- CD56dim CD16+
Volume of NK cells (CD56bright) | lutheal phase, day 20-28 in the menstrual cycle. The sample is collected at 9-10 AM and analysis is initiated within 60min.
  CD3- CD56bright CD16-
Volume of B-cells | lutheal phase, day 20-28 in the menstrual cycle. The sample is collected at 9-10 AM and analysis is initiated within 60min.
  CD3- CD19+ B cells
Volume of Th1 cells | lutheal phase, day 20-28 in the menstrual cycle. The sample is collected at 9-10 AM and analysis is initiated within 60min.
  CD3+CD4+ CXCR3+ CCR6- CCR10-
Volume of Th2 cells | lutheal phase, day 20-28 in the menstrual cycle. The sample is collected at 9-10 AM and analysis is initiated within 60min.
  CD3+CD4+ CCR4+ CCR6- CCR10-
Volume of Th17 cells | lutheal phase, day 20-28 in the menstrual cycle. The sample is collected at 9-10 AM and analysis is initiated within 60min.
  CD3+CD4+ CCR4+ CCR6+ CCR10-
Volume of Treg cells | lutheal phase, day 20-28 in the menstrual cycle. The sample is collected at 9-10 AM and analysis is initiated within 60min.
  CD25+CD127low

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Nørgaard-Pedersen, dr.med, Principal Investigator — Aalborg University Hospital, Denmark
Locations (1):
- • The Centre for Recurrent Pregnancy Loss of Western Denmark, Department of Obstetrics and Gynaecology, Aalborg University Hospital,, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
upon reasonable request
Supporting Information: Study Protocol, ICF, CSR
Time Frame: within 3 months
Access Criteria: upon reasonable request